CLINICAL TRIAL: NCT00896961
Title: Does Hypoxia Predict Radiation/Surgical Tumor Response/A Correlative Trial of EF5, an Agent for the Detection of Tumor Hypoxia
Brief Title: EF5 to Evaluate Tumor Hypoxia in Patients With High-Grade Soft Tissue Sarcoma or Mouth Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NCI-2012-02489; UPCC# 3300; CDR0000078671 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Stage I Adult Soft Tissue Sarcoma; Stage I Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage II Adult Soft Tissue Sarcoma; Stage II Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Adult Soft Tissue Sarcoma; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity
MeSH Terms: conditions — Sarcoma

ARMS (1):
- Observational (EF5) (Experimental): Approximately 24-48 hours prior to surgical resection or biopsy, patients receive EF5 IV over no more than 2½ hours. Tissue samples are analyzed by immunohistochemistry for EF5 binding. Blood samples are analyzed for genetic markers and cytokines associated with hypoxia and EF5 concentration.
  Interventions: Drug: EF5; Other: diagnostic laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: EF5
Other: diagnostic laboratory biomarker analysis
Other: pharmacological study
  Other Names: pharmacological studies

SUMMARY:
This laboratory study is using EF5 to evaluate tumor hypoxia in patients with high-grade soft tissue sarcoma or mouth cancer. Using the drug EF5 to measure the oxygen level in tumor cells may help in planning cancer treatment

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine biologically-relevant hypoxia by imaging and cellular analysis of EF5 binding in patients with high-grade soft tissue sarcoma of the trunk or extremity or squamous cell carcinoma of the oral cavity.

II. Determine the spatial relationships between EF5 binding and various tumor tissue markers, pathological processes, and serum plasminogen activator inhibitor-1 in these patients.

III. Correlate EF5 binding with Eppendorf electrode measurement and patient-related factors in these patients.

IV. Determine the adjusted and unadjusted associations between clinical outcome and optimal measures of EF5 binding, patient/tumor characteristics, and biological markers in these patients.

OUTLINE:

Approximately 24-48 hours prior to surgical resection or biopsy, patients receive EF5 IV over no more than 2½ hours. Tissue samples are analyzed by immunohistochemistry for EF5 binding. Blood samples are analyzed for genetic markers and cytokines associated with hypoxia and EF5 concentration.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high-grade soft tissue sarcoma (STS) of the trunk or extremity or squamous cell carcinoma of the oral cavity for which surgical biopsy or resection is standard initial therapy

  * Clinical imaging of mass that is likely to be STS or squamous cell carcinoma of the head and neck allowed if surgery is indicated prior to definitive diagnosis
* Planned resection and standard oncologic treatment
* No known distant metastatic disease
* ECOG 0-2
* WBC at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin less than 2.0 mg/dL
* Creatinine less than 2.0 mg/dL OR creatinine clearance at least 50 mL/min
* No significant cardiac condition that would preclude study compliance
* Weight no greater than 130 kg
* No grade III or IV peripheral neuropathy
* No other medical condition that would preclude study compliance
* Not pregnant or nursing
* Fertile patients must use effective contraception
* See Disease Characteristics
* No chemotherapy within 3 months before planned surgery
* Preoperative radiotherapy allowed for STS
* No radiotherapy within 3 months before planned surgery
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2001-08; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Time to locoregional recurrence in HNSCC patients | Time from study entry (EF5 administration) to locoregional recurrence, assessed up to 6 years
Time to distant metastasis in STS patients | Time from study entry (EF5 administration) to distant metastasis, assessed up to 6 years
How rapidly the STS recurred based on the original grade, time to recurrence and the degree of hypoxia in recurrent STS patients | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Michael Hahn, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States